CLINICAL TRIAL: NCT04102774
Title: Multicenter, Pragmatic, Randomized, Controlled Trial to Assess the Efficacy and Safety of Nocturnal Humidification Therapy in Patients With Bronchiectasis: the AIRVO-BX Study
Brief Title: Effect of AIRVO Heated Humidification in Bronchiectasis
Acronym: AIRVO-BX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Collaborators: ASST Fatebenefratelli Sacco (Other); Fondazione IRCCS Policlinico San Matteo di Pavia (Other); Ospedale Maggiore Di Trieste (Other); Azienda Ospedaliero-Universitaria di Modena (Other); Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other); Fondazione Salvatore Maugeri (Other); Università degli Studi di Ferrara (Other); Azienda Ospedaliero, Universitaria Pisana (Other); IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other); Ospedale San Paolo (Other); Universita degli Studi di Catania (Other); Azienda Ospedaliera di Padova (Other); University of Palermo (Other); Azienda Ospedaliero-Universitaria di Parma (Other); University of Foggia (Other); Monaldi Hospital (Other); Fondazione Don Carlo Gnocchi Onlus (Other); Ospedale San Donato (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AIRVO-BX
Record Dates: First submitted 2019-09-18; First posted 2019-09-25 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-05

CONDITIONS: Bronchiectasis Adult
Keywords: airway warm humidification; exacerbation; airway clearance

STUDY DESIGN:
Intervention Model Description: All the patients meeting inclusion/esclusion criteria will be enrolled and randomized into one of the two arms. The control arm will receive standard therapy. The treatment arm will receive standard therapy + long-term humidification therapy with myAIRVO2 at home overnight.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- myAIRVO2 (Experimental): Patients will receive a myAIRVO2 at home over-night with humidifier on top of standard therapy for bronchiectasis according to international guidelines (ERS 2017).
  Interventions: Device: Over-night treatment with myAIRVO2
- Control (No Intervention): Patients will receive standard therapy for bronchiectasis according to international guidelines (ERS 2017).

INTERVENTIONS:
Device: Over-night treatment with myAIRVO2 — Gas flow will be set between 20 and 30 l/min, according to patient's comfort, and administrated via nasal canula.
  Temperature will be set at 37°C. If the patient was already in nocturnal oxygen therapy FiO2 will be set according to the prescription.
  Arms: myAIRVO2

SUMMARY:
The aim of the study is to investigate whether long-term heated humidification therapy (AIRVO) administrated for 1 year over-night on top of standard therapy can reduce the number of exacerbations in adults with non-cystic fibrosis bronchiectasis.

DETAILED DESCRIPTION:
Bronchiectasis is a chronic condition characterized by an abnormal widened airways, mucus retention, cough, daily sputum, and frequent respiratory infections. The management of bronchiectasis includes prevention of exacerbations and lung infections along with airway clearance techniques.

Mucus composition and hydration are crucial to allow mucus transport along airways during respiratory physiotherapy.

Previous studies showed that long term humidification therapy increased airway clearance (Hasani et al. 2008) and reduced the number of exacerbations in patients with both bronchiectasis and Chronic Obstructive Pulmonary Disease (COPD) (Rea et al. 2010). myAIRVO2 system can deliver high-flow warm and humidified gases through a nasal cannula.

The aim of the present study to assess the effect of long-term use over-night of myAIRVO2 warm humidification in adults with bronchiectasis who experience at least 3 exacerbations/year still with optimized clinical and respiratory therapies.

In addition to their usual therapy, the treatment group will receive a myAIRVO2 humidifier at home deliver every day for one year over-night.

The gas flow setting will be set between 20 and 30 l/min based on patient preference, temperature will be 37°C and, for patients already in long-term oxygen therapy, FiO2 will be regulated according to patient's prescription.

The control group will continue to receive standard therapy for bronchiectasis according to international guidelines.

Patients will be screened during outpatient visits and, if they meet study criteria, they will be enrolled in the study. Once enrolled in the study, patients will be followed up every 3 months with 4 consecutive outpatient visits. The following endpoints will be assessed: exacerbations frequency, quality of life, pulmonary function and, for patients enrolled in the treatment group, myAIRVO2 use, and comfort.

Statistical analysis will be performed by Prof. Giovanni Sotgiu (University of Sassari - Italy).

ELIGIBILITY:
Inclusion Criteria:

* Radiological evidence of bronchiectasis evaluated through a CT-scan of the chest
* Daily sputum production
* Presence of at least 3 exacerbations requiring antibiotic therapy during the 12 months prior randomization
* Absence of exacerbations during the 28 days prior randomization
* Having the bronchiectasis management/therapy optimized according to international guidelines (ERS Polverino 2017) during the 12 months preceding randomization and no changes in therapy occurred during the 28 days prior randomization
* Airways clearance physiotherapy optimized and unchanged during the 12 months prior randomization
* Being able to use myAIRVO2 (assessed by study investigators)
* Given consent to inclusion in the study

Exclusion Criteria:

* Being enrolled in other intervention trials during the 12 months prior randomization
* COPD or asthma recognized as main diseases by the study investigator
* Active smoker or ex-smoker who underwent smoking cessation during the 4 weeks prior randomization
* Any other disease or medical condition diagnosed during the 3 months prior randomization which can affect patients' safety
* Long-term treatment with non-invasive ventilation (NIV)
* Long-term night treatment with continuous positive airway pressure (CPAP)
* Tracheostomy
* Major haemoptysis (more than 300ml or requiring embolization or requiring blood transfusion) during the 6 weeks prior randomization
* Cystic fibrosis
* Traction bronchiectasis in the context of pulmonary fibrosis
* Lung cancer in the last 5 years
* Use of drugs that can modify mucus liquid content including mannitol, Hypertoinc saline, DNase, NAC
* Changes in the rehabilitation/respiratory therapy program during the 28 days before randomization
* Pregnant and brest-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2025-01-31 (Actual); Study Completion 2025-01-31 (Actual)

PRIMARY OUTCOMES:
Pulmonary exacerbations | baseline - 12 months
  Number of pulmonary exacerbations

SECONDARY OUTCOMES:
Pulmonary exacerbations requiring hospitalization | baseline - 12 months
  Number of pulmonary exacerbations requiring hospitalization
Time to first pulmonary exacerbation | Up to 12 months. From date of randomization until the date of first documented pulmonary exacerbation
  Time occurring from the randomization to the first pulmonary exacerbation
Time to first hospitalization for exacerbation | Up to 12 months.From date of randomization until the date of first documented hospitalization for pulmonary exacerbation
  Time occurring from the randomization to the first exacerbation requiring hospitalization
Days with symptoms of exacerbation | baseline - 12 months
  Number of days the patient showed symptoms of exacerbation
Days of anibiotic treatment for exacerbation | baseline - 12 months
  Number of days of antibiotic treatment for exacerbation
Patients requiring de novo oxygen therapy | baseline - 12 months
  Number of patients starting de novo oxygen treatment
Quality-of-Life-Bronchiectasis Questionnaire, that measures health-related quality of life | baseline - 6 and 12 months
  We will measure changes in the score of Quality-of-Life-Bronchiectasis Questionnaire (QoL-B) completed by enrolled subjects at baseline and after 6 and 12 months.
  This disease-related questionnaire does not generate a total score, but a specific score for 8 different components: physical functioning domain, role functioning domain, vitality domain, emotional domain, social functioning domain, treatment burden domain, health perception domain and respiratory symptoms domain.
  For each component the scale range is 0 - 100, where higher scores correspond to better health status.
St.George Respiratory Questionnaire, that measures health-related quality of life | baseline - 6 and 12 months
  We will measure changes in the score of St.George Respiratory Questionnaire (SGRQ) completed by enrolled subjects at baseline and after 6 and 12 months.
  This questionnaire is structured into 3 main components: symptoms, activity and impacts.
  Scale range is 0-100, where lower scores correspond to the better health status.
  Each questionnaire response has a unique empirically derived "weight".
  Each component of the questionnaire is scored separately in three steps:
  i. The weights for all items with a positive responses are summed. ii The weights for missed items are deducted from the maximum possible weight for each component. The weights for all missed items are deducted from the maximum possible weight for the Total score.
  iii. The score is calculated by dividing the summed weights by the adjusted maximum possible weight for that component and expressing the result as a percentage The Total score is calculated in similar way.
Bronchiectasis Health Questionnaire, that measures health-related quality of life | baseline - 6 and 12 months
  We will measure changes in the score of Bronchiectasis Health Questionnaire (BHQ) completed by enrolled subjects at baseline and after 6 and 12 months.
  This disease-specific questionnaire generates a single total score. The maximum score is 79,42 and corresponds to a better health status, the minimum score is 26,77 and corresponds to a worse health status.
Leicester Cough Questionnaire, that measures health-related quality of life | baseline - 6 and 12 months
  We will measure changes in the score of Leicester Cough Questionnaire (LCQ) completed by enrolled subjects at baseline and after 6 and 12 months.
  This questionnaire consists of 19 items with a 7 point response scale. Each item is developed to assess impacts of cough on three main domains: physical, psychological and social.
  Scores are calculated as a mean of scores obtained for items of each domain (range 1 to 7).
  Total score is calculated by adding every single domain score (range 3-21). For both total and domains' scores higher values indicates better health status.
Pulmonary function as change in Forced Expiratory Volume in 1 Second (FEV1) | baseline - 6 and 12 months
  Change in FEV1, measured by spirometry
Pulmonary function as change in Forced Vital Capacity (FVC) | baseline - 6 and 12 months
  Change in FVC, measured by spirometry
Mortality | baseline - 12 months
  All-cause mortality
Mortality due to respiratory causes | baseline - 12 months
  Mortality rate caused by respiratory disease
Adverse events | baseline - 12 months
  Frequency and severity of adverse events
Non-use of AIRVO therapy | baseline - 12 months
  Frequency of permanent or temporary AIRVO therapy stopping

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Blasi, Prof, Principal Investigator — Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Locations (21):
- Italy (21):
  - IRCCS Humanitas Research Hospital, Department of Biomedical Sciences, Humanitas University,, Rozzano, Milano
  - Divisione di Pneumologia riabilitativa e Laboratorio di Citoimmunopatologia, Biochimica dell'apparato respiratorio, Istituti Clinici Scientifici Maugeri SpA - Società Benefit, Istituto di Ricovero e Cura a Carattere Scientifico, Veruno, Novara
  - Università degli Studi dell'Insubria e Istituti Clinici Scientifici Maugeri SpA - Società Benefit, Tradate, Varese
  - U.O.C Pneumologia e UTIP, Ospedale S. Donato, Arezzo
  - Dipartimento di Medicina Specialistica Diagnostica e Sperimentale, Alma Mater Studiorum, Università degli Studi di Bologna, Bologna
  - Dipartimento di Medicina Clinica e Sperimentale, U.O. di Fisiopatologia Respiratoria, Allergologia e Immunologia polmonare, Università degli Studi di Catania, Catania
  - Dipartimento di Scienze Mediche e Chirurgiche, Settore Malattie dell'Apparato Respiratorio, Università degli Studi di Foggia, Foggia
  - Department of Pathophysiology and Transplantation, University of Milan Internal Medicine Department, Respiratory Unit and Cystic Fibrosis Adult Center Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Dipartimento di Scienze biomediche e cliniche "Luigi Sacco" DIBIC, Università degli Studi di Milano, U.O.C Pneumologia, Ospedale L. Sacco - ASST Fatebenfratelli Sacco, Milan
  - Riabilitazione pneumologica, IRCCS Santa Maria nascente - fondazione don Gnocchi, Milan
  - U.O.C. Pneumologia, ASST- Santi Paolo e Carlo, Ospedale San Paolo, Dipartimento di Scienze della Salute, Università degli Studi di Milano, Milan
  - Struttura Complessa di Malattie dell'apparato Respiratorio e Centro delle Malattie Rare del Polmone, Dipartimento di Scienze Mediche e Chirurgiche Materno-Infantili e dell'Adulto, Università degli Studi di Modena e Reggio Emilia, Azienda Ospedaliero-Unive, Modena
  - U.O.C. Pneumologia SUN, Ospedale Monaldi, Napoli
  - Struttura Complessa di Fisiopatologia Respiratoria, Azienda Ospedaliera di Padova, Padua
  - Dipartimento Biomedico di Medicina Interna e Specialistica, Università degli Studi di Palermo, Palermo
  - Dipartimento di Medicina Clinica e Sperimentale, U.O.C. di Clinica Pneumologica, Azienda Ospedaliero-Universitaria di Parma, Parma
  - Dipartimento di Medicina Interna e Terapia Medica, Divisione di Malattie dell'Apparato Respiratorio, Fondazione IRCCS Policlinico San Matteo, Università degli Studi di Pavia, Pavia
  - U.O. di Riabilitazione Specialistica Pneumologica, Istituti Clinici Scientifici Maugeri SpA - Società Benefit, Istituto di Ricovero e Cura a Carattere Scientifico, Pavia
  - Unità Operativa Complessa di Pneumologia, Fondazione Policlinico Universitario A. Gemelli IRCCS, Università Cattolica del Sacro Cuore, Roma
  - U.O. di Riabilitazione Specialistica Pneumologica, Istituti Clinici Scientifici Maugeri SpA - Società Benefit, Istituto di Ricovero e Cura a Carattere Scientifico, Telese Terme
  - Struttura Complessa di Pneumologia, Ospedale di Cattinara, Azienda Sanitaria Universitaria Integrata di Trieste ex Azienda Ospedaliero-Universitaria "Ospedali Riuniti" di Tieste, Trieste

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hasani A, Chapman TH, McCool D, Smith RE, Dilworth JP, Agnew JE. Domiciliary humidification improves lung mucociliary clearance in patients with bronchiectasis. Chron Respir Dis. 2008;5(2):81-6. doi: 10.1177/1479972307087190. PMID 18539721
- [Background] Rea H, McAuley S, Jayaram L, Garrett J, Hockey H, Storey L, O'Donnell G, Haru L, Payton M, O'Donnell K. The clinical utility of long-term humidification therapy in chronic airway disease. Respir Med. 2010 Apr;104(4):525-33. doi: 10.1016/j.rmed.2009.12.016. Epub 2010 Feb 9. PMID 20144858
- [Background] Polverino E, Goeminne PC, McDonnell MJ, Aliberti S, Marshall SE, Loebinger MR, Murris M, Canton R, Torres A, Dimakou K, De Soyza A, Hill AT, Haworth CS, Vendrell M, Ringshausen FC, Subotic D, Wilson R, Vilaro J, Stallberg B, Welte T, Rohde G, Blasi F, Elborn S, Almagro M, Timothy A, Ruddy T, Tonia T, Rigau D, Chalmers JD. European Respiratory Society guidelines for the management of adult bronchiectasis. Eur Respir J. 2017 Sep 9;50(3):1700629. doi: 10.1183/13993003.00629-2017. Print 2017 Sep. PMID 28889110